CLINICAL TRIAL: NCT01329224
Title: Acetylsalicylic Acid in Outpatient Practice - Results From The Antiaggregation Monitoring (TAM) Registry
Brief Title: The Antiaggregation Monitoring (TAM) Registry
Acronym: TAM
Status: Completed | Type: Observational
Sponsor: Stephane Cook (Other)
Responsible Party: Sponsor-Investigator, Stephane Cook, Prof., University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Other Study IDs: 242/10A
Record Dates: First submitted 2011-03-30; First posted 2011-04-05 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2010-11

CONDITIONS: Aspirin Causing Adverse Effects in Therapeutic Use
Keywords: acetylsalicylic acid resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TAM patients: All consecutive patients under chronic ASA treatment (100mg/d) seen at our outpatient clinic.
  Interventions: Other: Measurement of platelet anti-aggregation

INTERVENTIONS:
Other: Measurement of platelet anti-aggregation — Whole blood impedance platelet aggregometry was performed with the Multiplate analyzer (Dynabyte, Munich, Germany) to test the response to ASA with arachidonic acid as the trigger.

SUMMARY:
The purpose of this study is to investigate the incidence of acetylsalicylic acid resistance (ASA-R) among patients under chronic acetylsalicylic acid(ASA) treatment seen at our outpatient clinic.

DETAILED DESCRIPTION:
Acetylsalicylic acid (ASA) resistance (R) is best defined as an ineffective inhibition of the platelet cyclooxygenase (COX)-1 pathway, and has been reported in 1 to 61 % of patients treated with ASA. Impaired response to ASA has been associated with an increased risk of ischemic events in patients with known coronary artery disease. We sought to investigate the incidence of ASA-R in clinical practice.

All consecutive patients under chronic ASA treatment (100mg/d) seen at our outpatient clinic were systematically included in the registry. All patients were on acetylsalicylic acid for CAD for at least 1 month. Patients were informed of ASA testing at start of consultation in the outpatient clinic. Eligible patients provided written informed consent. Peripheral venous blood samples were analyzed using the whole blood impedance platelet aggregometry Multiplate analyzer. The Multiplate analyzer device allows to measure platelet aggregation by the attachment of platelets to two silver coated copper electrodes leading to a rise of electrical resistance in the sample. The measurements are expressed as arbitrary aggregation units (AU) and the manufacturers defined cutoffs were used: normal values were 76-136 AU, partial antiaggregation was defined as ASA values between 31 and 75 AU and complete antiaggregation was defined as ASA values < 31 AU.

ELIGIBILITY:
Inclusion Criteria:

* patients under chronic ASA treatment for more then one month

Exclusion Criteria:

* concomitant use of nonsteroidal anti-inflammatory drugs (NSAIDs)
* thrombocytopenia
* thrombocytosis
* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients under chronic ASA treatment seen at our outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Whole blood impedance platelet aggregometry to assess acetylsalicylic acid resistance rates | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Cook, Prof, Principal Investigator — Fribourg University
Locations (1):
- Service de Cardiologie, Hôpital Cantonal Fribourg, Fribourg, Canton of Fribourg, Switzerland